CLINICAL TRIAL: NCT01405339
Title: The Effect of Budesonide Spray Via Mucosal Atomization Device on the Hypothalamic-Pituitary Axis
Brief Title: Budesonide Application Via Mucosal Atomization Device as a Treatment for Chronic Rhinosinusitis When Utilized as a Topical Nasal Steroid Spray
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, MD FRCSC FARS, Principal Investigator, Director of St Paul's Sinus Centre, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSMAD2011
Record Dates: First submitted 2011-07-26; First posted 2011-07-29 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide via MAD (Experimental): The current standard of care at St. Paul's Sinus Centre is to administer budesonide via the Mucosal Atomization Device (MAD). Its believed that MAD is a better device than the standard nasal lavage (Budesonide diluted in saline and delivered via Nasal Irrigation Bottle)because its fine mist and higher concentration enhances absorption and improves bioavailability.
  Interventions: Device: Mucosal Atomization Device (MAD)
- Budesonide via Sinus Rinse Bottle (Active Comparator): Budesonide via Sinus Rinse Bottle is the most commonly used delivery method.
  Interventions: Device: Budesonide via Nasal Syringe

INTERVENTIONS:
Device: Mucosal Atomization Device (MAD) — The use of pulmicort via MAD once a day for a total of 30 days.
  Arms: Budesonide via MAD
Device: Budesonide via Nasal Syringe — The use of budesonide via Sinus Irrigation Bottle will be once a day for 30 days.
  Arms: Budesonide via Sinus Rinse Bottle

SUMMARY:
Budesonide, a steroid subtype, has been used as an adjunctive treatment for chronic rhinosinusitis as a topical nasal steroid spray. The current standard of care at St. Paul's Sinus Centre is to administer budesonide via the Mucosal Atomization Device (MAD). It is believed that the MAD is a better device than the standard nasal lavage because its fine mist enhances absorption and improves bioavailability. No studies have been done to determine if enhanced absorption and improved bioavailability of budesonide via MAD could potentially affect the hypothalamic-pituitary-adrenal (HPA) axis, resulting in the suppression of our own body's production of natural steroids.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Diagnosed with CRS with or without polyps
* Awaiting for Functional Endoscopic Sinus Surgery
* Give consent on their own

Exclusion Criteria:

Concurrent or recent use (within the past 30 days) of systemic corticosteroids

* History of pituitary disease
* Morbid obesity (body mass index [calculated as weight in kilograms divided by height in meters squared]
* Concurrent or recent use of medications that accelerate the clearance of cortisol:

  o Such as dilantin, rifampin, amphetamines, or lithium carbonate
* Concurrent use of medications that interfere with the production of cortisol:

  o Such as ketoconazole, amphotericin B, bupropion, Echinacea, fluoroquinolones, itraconazole, licorice
* Use of oral contraception
* Use of female or male hormone therapy
* Known hypersensitivity to cortisol, corticotropin, or cosyntropin

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cosyntropin testing and blood work for quantification of plasma budesonide and plasma cortisol. | Participants will be followed for 30 days.

SECONDARY OUTCOMES:
SNOT-22 questionnaire to measure subjective perspective. | Participants will be followed for the duration of post op standard of care, an expected average of 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Amin R Javer, MD, FRCSC, FARS, Principal Investigator — St. Paul's Hospital, Canada
Locations (1):
- ENT Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Lund VJ, Black JH, Szabo LZ, Schrewelius C, Akerlund A. Efficacy and tolerability of budesonide aqueous nasal spray in chronic rhinosinusitis patients. Rhinology. 2004 Jun;42(2):57-62. PMID 15224630
- [Background] Sachanandani NS, Piccirillo JF, Kramper MA, Thawley SE, Vlahiotis A. The effect of nasally administered budesonide respules on adrenal cortex function in patients with chronic rhinosinusitis. Arch Otolaryngol Head Neck Surg. 2009 Mar;135(3):303-7. doi: 10.1001/archoto.2008.555. PMID 19289711
- [Background] Scott MB, Skoner DP. Short-term and long-term safety of budesonide inhalation suspension in infants and young children with persistent asthma. J Allergy Clin Immunol. 1999 Oct;104(4 Pt 2):200-9. doi: 10.1016/s0091-6749(99)70062-x. PMID 10518847
- [Background] Bhalla RK, Payton K, Wright ED. Safety of budesonide in saline sinonasal irrigations in the management of chronic rhinosinusitis with polyposis: lack of significant adrenal suppression. J Otolaryngol Head Neck Surg. 2008 Dec;37(6):821-5. PMID 19128710
- [Background] Kanowitz SJ, Batra PS, Citardi MJ. Topical budesonide via mucosal atomization device in refractory postoperative chronic rhinosinusitis. Otolaryngol Head Neck Surg. 2008 Jul;139(1):131-6. doi: 10.1016/j.otohns.2008.03.009. PMID 18585575
- [Derived] Thamboo A, Manji J, Szeitz A, Santos RD, Hathorn I, Gan EC, Alsaleh S, Javer AR. The safety and efficacy of short-term budesonide delivered via mucosal atomization device for chronic rhinosinusitis without nasal polyposis. Int Forum Allergy Rhinol. 2014 May;4(5):397-402. doi: 10.1002/alr.21280. Epub 2014 Jan 21. PMID 24449682